CLINICAL TRIAL: NCT03927339
Title: Aerobic Exercise and Knee Osteoarthritis
Brief Title: Do Obese Patients With Primary Knee Osteoarthritis Benefit From a Single Bout of Moderate Intensity Aerobic Exercise?
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: code R.18.04.137
Record Dates: First submitted 2019-04-16; First posted 2019-04-25 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2019-04

CONDITIONS: Knee Osteoarthriis and Oxidative Stress
Keywords: Osteoarthritis- Obesity- single aerobic exercise session

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pre and post excercise group
  Interventions: Diagnostic Test: pre and post excercise group

INTERVENTIONS:
Diagnostic Test: pre and post excercise group — Treadmill Training Protocol
  Each eligible participant in the patients group was then prospectively assigned to undergo exercise session of full-body-free weight treadmill training. Once the participants were prepped, they performed stretching for 5 min and slow walking for 3 min as a warm-up exercise before starting the training. Stretch was carried out similarly to all the subjects to quadriceps femoris and the hamstring. In the warm-up time period , it was enforced for 3 min at the speed of1 km/h. Then patients began the walking trials and walked at 1 to 1.34 m/s on an electric car treadmill (JACO fitness: JACO-212C).

SUMMARY:
Background: Obesity and degenerative joint disease are typically concomitant . Each are in the course of aerobic focus and excited inflammatory response. Exercise is taken into account a considerable treatment in rehabilitation of each conditions. nevertheless most of literature reported the good thing about regular exercise, whereas there's dearth regarding the consequence of base hit low to centrist usage session .

Objective:Hence, this report aimed to analyze the attainable effects of a single bout of moderate excercise in obese patients with KOA.

Methods:Thirty four rotund OA untrained semantic role and thirty age and sex matched healthy controls were registered during this sketch . OA patients were allotted to single session of low to moderate exercise on treadmill whereas controls remained unexercised. Perceived pain, GR activity, IL-6 , CRP, fasting blood glucose and lipid profile were assessed at baseline , once exercise and 24h after. Meanwhile, WOMAC score determined at baseline and once 24h.

DETAILED DESCRIPTION:
Study population:

This is an observational study a cohort of sedentary Egyptian patients included thirty four obese patients role diagnosed with primary human knee joint OA according to the criteria of the American College of Rheumatology (ACR)( 8).were selected from those attending the outpatient clinics of Rheumatology and Rehabilitation Department , Mansoura University (28 females and 6 males; mean age, 46.94 ± 10.84 years; trunk mass index, 40.91 ± 10.09 kg/m2). In addition, 30 healthy volunteers with no clinical and radiological evidence of OA(22 females and8 males; mean age,50.7 ±10.5 ; BMI 24.3±1.3)participated in the discipline .

Inclusion criteria: knee OA with obesity; sedentary with no previous education ; ability to understand and follow commands; and ability to walk independently.

Exclusion criteria: Medical conditions contraindicating moderate aerobic exercising (as determined through prescreening questions, i.e., cardiac or coronary artery disease as ischemic cardiomyopathy , chronic lung disease, asthma, uncontrolled hypertension), inability to exercise via treadmill(i.e. no neuromuscular or lower extremity conditions or any other medical contraindication that could prevent them from floor walking as upset affecting movement of the pelvic arch or pace , story of previous hip or knee operating room ,periarticular fractures, or lower limb injuries).History of recent reefer transmission or acute joint lighting .History of recent joint injection (steroid, hyaluronic acid , etc.) within 6 calendar week of study. Ingestion of antioxidant supplementation and the use of psychotropic agents.

Participants underwent bilateral AP standing x ray to verify the presence and degree of human knee OA. X-rays were marked exploitation the Kellgren and Lawrence (K/L) scale for knee OA severity(9).Subjects with picture taking knee OA of KL grade ≥2 in a minimum of one knee were listed. The grading of the worst affected knee in every patient was used for knowledge analysis.

Physical examinations including age and body mass index (BMI) were obtained at the same visits at which radiographs were obtained. Western Ontario and McMaster Universities Arthritis Index (WOMAC) scores of the OA patients were collected (10).

Treadmill Training Protocol

Each eligible participant in the patients group was then prospectively assigned to undergo exercise session of full-body-free weight treadmill training. Once the participants were prepped, they performed stretching for 5 min and slow walking for 3 min as a warm-up exercise before starting the training. Stretch was carried out similarly to all the subjects to quadriceps femoris and the hamstring. In the warm-up time period , it was enforced for 3 min at the speed of1 km/h. Then patients began the walking trials and walked at 1 to 1.34 m/s on an electric car treadmill (JACO fitness: JACO-212C).

Exercise intensity

For the purpose of this study, Metabolic Equivalents (METs) and Rate of Perceived Exertion (RPE) were used as guidelines to determine exercise intensity. Moderate aerobic exercise has been objectively defined as activity that generates energy expenditure of 3.0 to 6.0 (METs) (11).

To determine the intensity, time and frequency of exercise, it was set at low to moderate, that is between 40% and 60% of the maximum heart rate, from 12 to 14 rating of RPE. In addition, each subject was shown the 15 point Borg Rating of Perceived Exertion scale and instructed in its use. The RPE scale was mounted on the wall in front of the treadmill and easily visible to the subjects. Exercise instructions and measurements of associated Metabolic Equivalents (METs) were determined based upon previous studies which determined that walking on a level surface at 3.0 MPH equates to 3.3 METs and walking at 4.5 MPH generates 6.3 METs(12).

Participants walked at a pace of 2.5 to 3.0 MPH on a treadmill with zero incline for 30 min and they were instructed to walk at a pace that neither caused pain nor increased symptoms (13).

To minimize pain that may occur due to treadmill exercise, 5 min rest were allowed after 15 min of exercise. In the control group, the subjects remained at rest.

The present study was conducted in agreement with the guidelines of the Declaration of Helsinki. Written informed consent was received from every patient and healthy subject before participating in the study. This study was approved by the Institutional Research Board of the Faculty of Medicine, Mansoura University code R.18.04.137

Laboratory assays:

Blood samples were drawn before and once exercise (within 0.5 h once exercise,and at 24 h). All organic chemistry measurements were performed on frozen plasma samples obtained by activity of freshly drawn blood (3000 × g for 20minutes at 4∘C) and consequent storage at -70∘C. Blood macromolecule profiles, together with total cholesterol (TC), HDL cholesterol (HDL-C), calculated LDL cholesterol(LDL-C), and triglycerides (TG) concentrations were determined by protein assays., further as abstinence blood sugar level.

IL-6, CRP Serum concentrations of IL-6 were determined using sandwich high sensitivity ELISA kit for quantitative detection of human IL-6 according to manufacturer's protocol (Boster Immunoleader by Boster Biological Technology Co. Inc.). Detection of serum CRP was performed by Solid Phase Sandwich ELISA according to manufacturer's instructions (Quantikine Human CRP Immunoassay, R&D systems)

Glutathione reductase assay:

Spectrophotometric determination of GR activity in the serum was measured as described by Calberg and Mannervic (14) using commercially available Glutathione Reductase Assay Kit(Sigma chemical company, St Louis, Missouri, USA). Glutathione reductase catalyzes the reduction of GSSG by oxidizing NADPH to NADP+. The decrease in absorbance was measured at 340.

ELIGIBILITY:
Inclusion Criteria:

* : knee OA with obesity; sedentary with no previous education ; ability to understand and follow commands; and ability to walk independently.

Exclusion Criteria:

* Medical conditions contraindicating moderate aerobic exercising (as determined through prescreening questions, i.e., cardiac or coronary artery disease as ischemic cardiomyopathy , chronic lung disease, asthma, uncontrolled hypertension), inability to exercise via treadmill(i.e. no neuromuscular or lower extremity conditions or any other medical contraindication that could prevent them from floor walking as upset affecting movement of the pelvic arch or pace , story of previous hip or knee operating room ,periarticular fractures, or lower limb injuries).History of recent reefer transmission or acute joint lighting .History of recent joint injection (steroid, hyaluronic acid , etc.) within 6 calendar week of study. Ingestion of antioxidant supplementation and the use of psychotropic agents.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: a cohort of egyptian patients suffering from obesity and knee osteoarthritis
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2019-06-29 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
change in degree of pain from base line | assessed immediately before excercise, 10 minutes after excercise and 24 hours after excercise
  1-Pain Visual Analogue Scale: The VAS-pain score is composed of a continuous horizontal line. This line is 100 mm in length. To measure the intensity of pain, the score is anchored by (0 score = no pain) at one end and (100 score = worst imaginable pain) on the other end. The patient places a mark to the VAS line at the point which represents the intensity of his pain(1
CHange in function from base line | Assessed before excercise immediately,10 minutes after, excercise,24 hours after excercise
  Western Ontario and McMaster Universities Arthritis Index (WOMAC) scores of the OA patients were collected (10).
  Scores from the Western Ontario and Mc-Master University (WOMAC) OA index were used to assess pain, stiffness and function in OA patients [11]. Total WOMAC is the sum of 3 subscales scores. High WOMAC score indicates more pain and stiffness and severe functional limitation.

SECONDARY OUTCOMES:
CHANGE INserum IL6 FROM BASE LINE, | assessed immediately before excercise, 10 minutesafter excercise,and 24 hours after excercise
  Serum concentrations of IL-6 were determined using sandwich high sensitivity ELISA kit for quantitative detection of human IL-6 according to manufacturer's protocol (Boster Immunoleader by Boster Biological Technology Co. Inc.)
change in serum C REACTIVE PROTEIN from base line | assessed immediately before excercise, 10 minutesafter excercise,and 24 hours after excercise
  Detection of serum CRP was performed by Solid Phase Sandwich ELISA according to manufacturer's instructions (Quantikine Human CRP Immunoassay, R&D systems)
change inSERUM LIPID PROFILE from base line | assessed immediately before excercise, 10 minutesafter excercise,and 24 hours after excercise
  Blood macromolecule profiles, together with total cholesterol (TC), HDL cholesterol (HDL-C), calculated LDL cholesterol(LDL-C), and triglycerides (TG) concentrations were determined by protein assays.,
change in serum Glutathione reductase assay: from base line | assessed immediately before excercise, 10 minutesafter excercise,and 24 hours after excercise
  Spectrophotometric determination of GR activity in the serum was measured as described by Calberg and Mannervic (14) using commercially available Glutathione Reductase Assay Kit(Sigma chemical company, St Louis, Missouri, USA). Glutathione reductase catalyzes the reduction of GSSG by oxidizing NADPH to NADP+. The decrease in absorbance was measured at 340.

CONTACTS AND LOCATIONS:
Locations (1):
- Reham Magdy Shaat, Al Mansurah, Dakahlia Provence, Egypt